CLINICAL TRIAL: NCT00272805
Title: Prospective, Randomized, Controlled Assessment of Once-Daily Controlled Release COREG CR vs Twice-Daily COREG Immediate Release(IR)on Measures of Compliance and Quality of Life in Patients With Heart Failure and Left Ventricular Systolic Dysfunction
Brief Title: Drug Compliance and Quality of Life in Patients With Heart Failure Dosed With Either Once-daily or Twice-daily Coreg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cardiovascular Clinical Sciences Inc (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCS 2005-001; CASPER
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; left ventricular systolic dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Carvedilol

INTERVENTIONS:
Drug: carvedilol

SUMMARY:
The purpose of this study is to compare dosing compliance between study patients taking controlled release carvedilol once a day, and study patients taking immediate release carvedilol (Coreg) twice a day.

DETAILED DESCRIPTION:
Study Further Study Details:

Primary outcome: pill-taking compliance (total doses taken versus total doses prescribed)

Expected Total Enrollment: 400 subjects at 56 study sites in the U.S.

Study Start: October 2005

This is a 5-month double-blind treatment study of male and female subjects with stable mild-to-severe chronic heart failure and with left ventricular dysfunction with symptoms of heart failure.

Eligibility:

Must be stable on treatment with Coreg IR at a standard dose: 6.25, 12.5, 25 mg twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read English
* Stable symptoms of mild to severe heart failure
* Stable medical regimen for heart failure
* On a stable dose of Coreg for at least 2 months
* LVEF ≤40% within the previous 24 months

Exclusion Criteria:

* Uncorrected obstructive or regurgitant valve disease
* Complex congenital heart disease
* Recent ICD or pacemaker placement
* Recent coronary artery bypass surgery or stroke
* Candidate for heart transplanct within 5 months of study start
* Present or planned use of MAO inhibitors, alfpha-blockers, combined alpha-beta blockers, any Class I/II anti-arrythmnic agents, (amiodarone may be used if ≤ 200mg/day). Use of intravenous vasodilator/inotropic agents.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Dosing compliance: pill taking total taken vs number prescribed

SECONDARY OUTCOMES:
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: James E. Udelson, M.D., Principal Investigator — Cardiovascular Clinical Studies, Inc.
Locations (54):
- United States (54):
  - The Heart Group, Mobile, Alabama
  - Radiant Research, Sierra Vista, Arizona
  - Cardiology Consultants of Orange County, Anaheim, California
  - Access Clinical Trials, Beverly Hills, California
  - Cardiovascular Consultants Medical Group, Oakland, California
  - San Diego Cardiac Center, San Diego, California
  - Northern California Medical Associates, Santa Rosa, California
  - Radiant Research, Santa Rosa, California
  - Cardiovascular Consultants Medical Group, Walnut Creek, California
  - Heart Center of the Rockies, Fort Collins, Colorado
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - NextPhase Clinical Trials, Miami, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - The Heart and Vascular Institute of Florida, St. Petersburg, Florida
  - Cardiac Disease Specialists, Atlanta, Georgia
  - CVMS Research Institute of Augusta, Augusta, Georgia
  - Georgia Heart Specialists, Covington, Georgia
  - Idaho Cardiology Associates, Boise, Idaho
  - North Shore Cardiologists, Bannockburn, Illinois
  - Midwest Heart Foundation, Lombard, Illinois
  - Illinois Heart and Lung Research Center, Normal, Illinois
  - The Care Group, Indianapolis, Indiana
  - Clinical Trials Management, Metairie, Louisiana
  - Androscoggin Cardiology Associates-Research, Auburn, Maine
  - Maine Cardiology Associates, S.Portland, Maine
  - Cardiovascular Consultants of Maine, Scarborough, Maine
  - Primary Care Cardiology Research, Ayer, Massachusetts
  - Lahey Clinic Cardiology, Burlington, Massachusetts
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - Lovelace Scientific Resources, Las Vegas, Nevada
  - Associated Cardiovascular Consultants, Cherry Hill, New Jersey
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - Albany Associates in Cardiology, Albany, New York
  - Cardiovascular Medical Associates, Garden City, New York
  - MidValley Cardiology, Kingston, New York
  - New York University Medical School, New York, New York
  - South Bay Cardiovascular Associates, West Islip, New York
  - Alamance Regional Medical Center, Burlington, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - The Dayton Heart Center, Dayton, Ohio
  - North Ohio Research Ltd., Lorain, Ohio
  - North Ohio Research Ltd., Sandusky, Ohio
  - Blue Stem Cardiology, Bartlesville, Oklahoma
  - Cardiovascular Consultants of Oregon, Corvallis, Oregon
  - Oregon Medical Group Clinical Research, Eugene, Oregon
  - Guthrie Clinic Ltd., Sayre, Pennsylvania
  - Rhode Island Heart Failure Center, Providence, Rhode Island
  - DCOL Center for Clinical Research, Longview, Texas
  - LDS Hospital Cardiovascular Research, Salt Lake City, Utah
  - Arrythmia Center for Southern Wisconsin, Elkhorn, Wisconsin

REFERENCES:
- [Derived] Udelson JE, Pressler SJ, Sackner-Bernstein J, Massaro J, Ordronneau P, Lukas MA, Hauptman PJ. Adherence with once daily versus twice daily carvedilol in patients with heart failure: the Compliance And Quality of Life Study Comparing Once-Daily Controlled-Release Carvedilol CR and Twice-Daily Immediate-Release Carvedilol IR in Patients with Heart Failure (CASPER) Trial. J Card Fail. 2009 Jun;15(5):385-93. doi: 10.1016/j.cardfail.2008.12.010. Epub 2009 Feb 12. PMID 19477398